CLINICAL TRIAL: NCT01414738
Title: Phase II Trial of Hippocampal-Avoiding Whole Brain Irradiation With Simultaneous Integrated Boost for Treatment of Brain Metastases
Brief Title: Hippocampal-Avoiding Whole Brain Irradiation With Simultaneous Integrated Boost for Treatment of Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Timmerman, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 042011-050
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2020-03

CONDITIONS: Brain Neoplasms, Adult, Malignant
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation (Experimental): Whole-Brain Radiotherapy
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Hippocampal-Avoiding Whole Brain Irradiation with Simultaneous Integrated Boost

SUMMARY:
The investigators hypothesize that avoidance of the hippocampal region with WBRT (Whole-Brain Radiotherapy ) may delay or reduce the onset, frequency, and/or severity of NCF (neurocognitive function) decline, as measured with clinical neurocognitive tools.

DETAILED DESCRIPTION:
We propose to use conformal avoidance of the hippocampal region during whole brain radiotherapy to reduce the dose to the hippocampi, thereby putatively limiting the radiation-induced inflammation of the hippocampal region and subsequent alteration of the microenvironment of the neural progenitor cells

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically (histologically or cytologically) proven diagnosis of a non-hematopoietic malignancy other than small cell lung cancer and germ cell malignancy.. Direct biopsy of CNS (central nervous system) lesions is not necessarily required although could constitute an allowed site of tissue confirmation as medically prudent. Patients who have been disease free for more than 5 years prior to the appearance of CNS metastases should undergo repeat biopsy of either a systemic metastasis or the CNS metastases to confirm the recurrent malignancy.
2. Patients with measurable brain metastasis outside a 5-mm margin around either hippocampus
3. Patients with measurable brain metastasis who have not been or will not be treated with SRS (stereotactic radiosurgery ) or surgical resection (Note: These treatment options are only permitted at relapse)
4. History/physical examination within 28 days prior to registration
5. Patients must fall into RTOG (Radiation Therapy Oncology Group) recursive partitioning analysis (RPA) class I or II
6. Patients must have a life expectancy of at least 4 months.
7. Age ≥ 18 years
8. Karnofsky performance status ≥ 70
9. Patients must provide study-specific informed consent prior to study entry
10. Women of childbearing potential and male participants must practice adequate contraception
11. Women of childbearing potential must have a negative, qualitative serum pregnancy test ≤2 weeks prior to study entry

Exclusion Criteria:

1. Patients with greater than 9 discrete metastases on MRI.
2. Patients with leptomeningeal metastases
3. Patients with measurable brain metastasis not resulting from small cell lung cancer and germ cell malignancy
4. Plan for chemotherapy or targeted therapies during WBRT or over the subsequent 7 days
5. Contraindication to MR (Magnetic resonance) imaging such as implanted metal devices or foreign bodies, severe claustrophobia AND patients unable to receive gadolinium contrast agents
6. Serum creatinine > 1.4 mg/dl ≤ 28 days prior to study entry
7. Prior radiation therapy to the brain
8. Patients planning to undergo radiosurgery to any CNS lesion OR patients planning to have surgical resection of ALL of their CNS lesions

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10-18 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Timmerman, MD, Principal Investigator — UT Southwestern Medical Center Dallas
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation
Started (1 patient did not initiate treatment) | 49
Follow-up (3 Months) | 18
Follow-up (6 Months) | 8
Follow-up (9 Months) | 5
Completed | 5
Not Completed | 44
Not completed — Death | 26
Not completed — Refused testing | 5
Not completed — Lost to Follow-up | 2
Not completed — Refused, disease progression | 8
Not completed — (Unknown) NOS (Not Otherwise Specified) | 3

BASELINE CHARACTERISTICS:
Arm/Group | Radiation
Number analyzed (Participants) | 49
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [54 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31
  African American | 11
  Other | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in *Delayed* Recall Score by Hopkins Verbal Learning Test-Revised (HVLT-R DR) Score
Description: The HVLT-R is a validated test to assess neurocognitive function and it incorporates 6 different forms, each including 12 nouns (targets) with 4 words drawn from 3 semantic categories.
  *Delayed*recall was measured by recalling the 12 targets after a 20-minute delay.
  1 point is awarded for each successfully recalled target. There is no range- recalling more is more memory.
  Mean change was calculated by the following formula: 100*(3 month - baseline) / baseline
Time Frame: Baseline, 3 months
Population: Complete case analysis was done for this and 1 participant who missed the test was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage difference
Arm/Group | Radiation
Number analyzed (Participants) | 17
percentage difference | -10.6 (50.4)

2. Secondary Outcome: Mean Change in *Immediate* Recall Score by Hopkins Verbal Learning Test-Revised (HVLT-R)
Description: The HVLT-R is a validated test to assess neurocognitive function and it incorporates 6 different forms, each including 12 nouns (targets) with 4 words drawn from 3 semantic categories.
  *Immediate* recall was measured by memorizing a list of 12 targets for 3 consecutive trials.
  1 point is awarded for each successfully recalled target. There is no range- recalling more is more memory.
  Mean change was calculated by the following formula: 100*(3 month - baseline) / baseline
Time Frame: Baseline, at 3 months
Population: Complete case analysis was done for this and 1 participant who missed the test was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage difference
Arm/Group | Radiation
Number analyzed (Participants) | 17
percentage difference | 39.6 (129.4)

3. Secondary Outcome: Mean Change in *Delayed Recognition* Score by Hopkins Verbal Learning Test-Revised (HVLT-R)
Description: The HVLT-R is a validated test to assess neurocognitive function and it incorporates 6 different forms, each including 12 nouns (targets) with 4 words drawn from 3 semantic categories.
  *Delayed recognition* was measured by using recognition discrimination index.
  1 point is awarded for each successfully recalled target. There is no range- recalling more is more memory.
  Mean change was calculated by the following formula: 100*(3 month - baseline) / baseline
Time Frame: Baseline, 3 months
Population: Complete case analysis was done for this and 1 participant who missed the test was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage difference
Arm/Group | Radiation
Number analyzed (Participants) | 17
percentage difference | -0.4 (19.9)

4. Secondary Outcome: Mean Change in Neurocognitive Function as Measured by Controlled Word Association Test
Description: Controlled Word Association Test (COWAT) is used to assess language and executive/frontal skills. The patient produces as many words as possible in 1 min. (each) for a specific letter (C, F, L or P, R, W). Requires about 5 min to complete.
  1 point is awarded for each word produced. Mean change was calculated by the following formula: 100*(3 month - baseline) / baseline
Time Frame: Baseline, at 3 months
Population: Complete case analysis was done for this and 1 participant who missed the test was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage difference
Arm/Group | Radiation
Number analyzed (Participants) | 17
percentage difference | 3.7 (40.0)

5. Secondary Outcome: Mean Change in Trail Making Test (TMT- A) Score
Description: Trail Making Test (TMT) is a measure of visuospatial scanning, attention, sequencing, and speed and executive function. Patients must "connect the dots" either in a numbered sequence or alternating letters and numbers.
  The TMT has two parts that are referred to as the Trail Making Test Part A and the Trail Making Test Part B.
  In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order.
  Possible score ranges from 0-3 minutes with higher score (more seconds/minutes) indicating significant cognitive impairment.
  Mean change was calculated by the following formula: 100*(3 month - baseline) / baseline
Time Frame: Baseline, at 3 months
Population: Complete case analysis was done for this and 2 participants who missed the test were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage difference
Arm/Group | Radiation
Number analyzed (Participants) | 16
percentage difference | 17.7 (86.6)

6. Secondary Outcome: Mean Change in Trail Making Test (TMT- B) Score
Description: Trail Making Test (TMT) is a measure of visuospatial scanning, attention, sequencing, and speed and executive function. Patients must "connect the dots" either in a numbered sequence or alternating letters and numbers.
  The TMT has two parts that are referred to as the Trail Making Test Part A and the Trail Making Test Part B.
  In Part B, the circles include both numbers (1 - 13) and letters (A - L). Possible score ranges from 0-5 minutes with higher score (more seconds/minutes) indicating significant cognitive impairment.
Time Frame: Baseline, at 3 months
Population: Complete case analysis was done for this and 4 participants who missed the test were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage difference
Arm/Group | Radiation
Number analyzed (Participants) | 14
percentage difference | 12.0 (34.9)

7. Secondary Outcome: Mean Change in Cognitive Function as Measured by Medical Outcomes Scale (MOS)
Description: Medical Outcomes Scale (MOS) assess cognitive function with possible score range from 0-100, with higher scores indicating better outcome.
  Mean change was calculated by the following formula: 100*(3 month - baseline) / baseline
Time Frame: Baseline, at 3 months
Population: Complete case analysis was done for this and 1 participant who missed the test was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage difference
Arm/Group | Radiation
Number analyzed (Participants) | 17
percentage difference | 3.2 (18.2)

8. Secondary Outcome: Mean Change in Cognitive Function as Measured by Mini-Mental Status Examination (MMSE)
Description: Mini-Mental Status Examination (MMSE) is a brief, standardized tool to grade patients' global cognitive function. Possible scores range from 0-30, with lower score indicating severe cognitive impairment.
  Mean change was calculated by the following formula: 100*(3 month - baseline) / baseline
Time Frame: Baseline, at 3 months
Population: Complete case analysis was done for this and 1 participant who missed the test was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage difference
Arm/Group | Radiation
Number analyzed (Participants) | 17
percentage difference | -0.1 (7.0)

9. Secondary Outcome: Mean Change in Relative Fatigue as Measured by Multidimensional Fatigue Inventory (MFI-20) Scores
Description: The MFI-20 is a multidimensional, self-reporting instrument designed to measure fatigue. It covers the following dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. Possible subscore ranges from 4 to 20 is reported for each dimension, with 20 corresponding to maximal fatigue.
Time Frame: Baseline, 3 months
Population: Complete case analysis was done for this and 2 participants who missed the test were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage difference
Arm/Group | Radiation
Number analyzed (Participants) | 16
percentage difference | 6.6 (32.2)

10. Secondary Outcome: Cumulative Incidence of Local Failure
Description: Cumulative incidence of local failure, defined as tumor recurrence . Percent local failure at 1 year.
  The Cox proportional hazards regression model will be used to evaluate Cumulative incidence of local failure.
  This is to evaluate local control of brain metastases treated with integrated boost.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: hazard (probability) of tumor recurrence
Arm/Group | Radiation
Number analyzed (Participants) | 49
hazard (probability) of tumor recurrence | 8.8 [2.7 to 19.6]

11. Secondary Outcome: Cumulative Incidence of Intracranial Failure
Description: Cumulative incidence of intracranial failure was estimated by the Cox proportional hazards regression model.
  Intracranial failure is any failure in the brain.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: hazard (probability) of tumor recurrence
Arm/Group | Radiation
Number analyzed (Participants) | 49
hazard (probability) of tumor recurrence | 21.3 [10.7 to 34.2]

12. Secondary Outcome: Percentage of Participants With Local Failures Within the Region of Brain Within the CTV Receiving 20 Gy
Description: Percentage of participants with local failures within the region of brain within the CTV (Clinical Target Volume ) receiving 20 Gy
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Radiation
Number analyzed (Participants) | 49
percentage of participants | 10.5

13. Secondary Outcome: Number of Participants With Recurrence in the Hippocampus
Description: Recurrence in the hippocampus was noted after hippocampal-sparing whole brain irradiation with simultaneous integrated boost (HSIB-WBRT)
Time Frame: 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation
Number analyzed (Participants) | 49
Participants | 1

14. Secondary Outcome: Median Progression Free Survival
Description: Tumor progression is measured radiographically. The Kaplan-Meier estimator was used to determine the median time to death for this patient population.
Time Frame: 39 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation
Number analyzed (Participants) | 49
months | 2.9 [1.5 to 4.0]

15. Secondary Outcome: Median Overall Survival.
Description: Overall survival is measured by the Kaplan-Meier estimator used to determine the median overall survival for this patient population.
Time Frame: 39 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation
Number analyzed (Participants) | 49
months | 9 [4.07 to 14.87]

16. Secondary Outcome: Number of Adverse Events Grade 3 or Higher Based on CTCAE (Common Terminology Criteria for Adverse Events) Criteria.
Description: The adverse event (AE) including any adverse event would be assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: From start of treatment up to 39 months
Measure: Number; unit: events
Arm/Group | Radiation
Number analyzed (Participants) | 49
events | 3

17. Secondary Outcome: Health-related Quality of Life as Assessed by the Functional Assessment of Cancer Therapy With Brain Subscale (FACT-BR)
Description: Quality of life will be assessed using the Functional Assessment of Cancer Therapy with Brain Subscale (FACT-BR). The FACT-BR is a multidimensional, self-report quality of life instrument specifically designed and validated for use with brain malignancy patients. It is written at the 4th grade reading level and can be completed in 5-10 minutes with little or no assistance in patients who are not neurologically incapacitated. It measures quality of life related to symptoms or problems across 5 scales: physical well-being (7 items); social/family well-being (7 items);emotional well-being (6 items); functional well-being (7 items); and concerns relevant to patients with brain tumors (23 items).
  Items are rated on a 5-point scale (0-5): 0-"not at all", 1- "a little bit", 2-"somewhat", 3-"quite a bit" and 4-"very much", with HIGHER scores indicating a better quality of life.
Time Frame: 39 months
Population: This data was not collected as we were no longer interested in collecting this.
Arm/Group | Radiation
Number analyzed (Participants) | 0

18. Secondary Outcome: Health-related Quality of Life as Assessed by Euroqol EQ-5D
Description: The EQ (Euroqol)-5D (5 Dimension) health related quality of life questionnaire is a standardized instrument for use as a measure of health outcome.
  Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status. . The US version of the EQ-5D will be used, to enable mapping of general HR-QoL (Health-related quality of life) scores from EQ-5D scores into health state utility scores (ranging from 0 to 1) for the US population.
  Possible scores range from 0 to 1, with HIGHER scores indicating a better quality of life.
Time Frame: 39 months
Population: This data was not collected as we were no longer interested in collecting this.
Arm/Group | Radiation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 39 months
Arm/Group | Radiation
All-Cause Mortality (participants affected / at risk) | 26/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 13/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation (N=49)
Alopecia (Skin and subcutaneous tissue disorders) | 4
Fatigue (Nervous system disorders) | 13
Anorexia (Metabolism and nutrition disorders) | 2
Aphasia (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dizziness (General disorders) | 2
Dysarthria (Nervous system disorders) | 1
Edema face (Blood and lymphatic system disorders) | 1
Gait disturbance (Nervous system disorders) | 1
Headache (General disorders) | 10
Hearing loss (Ear and labyrinth disorders) | 1
Insomnia (General disorders) | 1
Nausea (General disorders) | 10
Seizures (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 2

LIMITATIONS AND CAVEATS:
SAE (Serious Adverse Events) were not analyzed on a per patient basis and hence reported as '0' within the AE module.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT01414738/Prot_SAP_000.pdf